CLINICAL TRIAL: NCT05367232
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of ICP-033 in Patients With Solid Tumors
Brief Title: A Study of ICP-033 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00701
Record Dates: First submitted 2022-04-24; First posted 2022-05-10 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Patients With Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-033 Dose Escalation (Experimental): Drug: ICP-033 tablet Administered orally，once a day，every 28 days is a cycle.
  Interventions: Drug: ICP-033 tablet

INTERVENTIONS:
Drug: ICP-033 tablet — Administered orally, once a day, 28 days per cycle

SUMMARY:
A Dose finding Study to Evaluate the Safety, Tolerability and Pharmacokinetics and Preliminary Anti-Tumor Activity of ICP-033 Tablets in Patients with Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
2. Patients with histologically confirmed locally advanced unresectable or metastatic solid tumors;
3. At least one measurable lesion according to RECIST 1.1.

Exclusion Criteria:

1. Pregnant and lactating women, or women planning to become pregnant during the study through at least 6 months after the last dose of study drug.
2. Patients with unstable primary central nervous system (CNS) tumors or CNS metastases.
3. Patients who have active or history of interstitial lung disease or noninfectious pneumonia.
4. Patients with QTc > 450 ms in males and > 470 ms in females on ECG at screening, or other clinically significant abnormalities in the ECG at the discretion of the investigator.
5. Patient with the Medication history and surgical history as stated in the protocol
6. Those who are unsuitable for blood collection or contraindicated for blood collection.
7. Other conditions considered unsuitable for participation in this trial at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse event (AE) of ICP-033 assessed by NCI-CTCAE V5.0. | through study completion, an average of 2 years
  To assess the safety and tolerability of ICP-033 in patients with advanced solid tumors.
Dose-Limiting Toxicities (DLTs) | through study completion, an average of 2 years
  To assess the safety and tolerability of ICP-033 in patients with advanced solid tumors.
Maximum tolerated dose (MTD) | through study completion, an average of 2 years
  To assess the safety and tolerability of ICP-033 in patients with advanced solid tumors.
Recommended phase II dose (RP2D) | through study completion, an average of 2 years

SECONDARY OUTCOMES:
The maximum plasma concentration observed (Cmax) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-033 in patients with solid tumors.
Time of maximum observed plasma concentration (Tmax) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-033 in patients with solid tumors.
Elimination half-life (t1/2) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-033 in patients with solid tumors.
Area under plasma concentration-time curve (AUC0-t and AUC0-∞) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-033 in patients with solid tumors.
Apparent clearance (CL/F) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-033 in patients with solid tumors.
Apparent volume of distribution (Vz/F) | through study completion, an average of 2 years
  To evaluate the pharmacokinetic (PK) characteristics of ICP-033 in patients with solid tumors.
The objective response rate (ORR) | through study completion, an average of 2 years
  To evaluate the preliminary anti-tumor activity of ICP-033.
Duration of response (DoR) | through study completion, an average of 2 years
  To evaluate the preliminary anti-tumor activity of ICP-033.
Progression-free survival (PFS) | through study completion, an average of 2 years
  To evaluate the preliminary anti-tumor activity of ICP-033.
Overall survival (OS) | through study completion, an average of 2 years
  To evaluate the preliminary anti-tumor activity of ICP-033.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Bi, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Sichuan, Chengdu, China